CLINICAL TRIAL: NCT03799666
Title: (Re)Vitalizing Pulmonary Rehabilitation
Brief Title: (Re)Vitalizing Pulmonary Rehabilitation for Patients With Chronic Respiratory Diseases
Acronym: 3R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Alda Sofia Pires de Dias Marques, Senior Lecturer, Aveiro University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAICT-POL/23926/2016
Record Dates: First submitted 2018-12-14; First posted 2019-01-10 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Chronic Respiratory Disease
Keywords: Pulmonary rehabilitation; Community-based; Chronic Respiratory Diseases; Cost-benefit analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary Rehabilitation Group (Experimental): Patients will participate in a 12-week community-based pulmonary rehabilitation programme.
  Interventions: Other: Pulmonary Rehabilitation
- Standard Care Group (Active Comparator): Patients will continue to receive the standard care, which means the daily medication prescribed by the pshysician from the primary care centre team.
  Interventions: Other: Daily medication

INTERVENTIONS:
Other: Pulmonary Rehabilitation — Patients will be treated with daily medication prescribed by the physician. Additionally patients will participate in a 12-w.eek community-based pulmonary rehabilitation programme, with two exercise training sessions per week and six psycho-education sessions, managed by a multidisciplinary team, once every two weeks. Patient's families will be invited to participate in the psychoeducational component
  Arms: Pulmonary Rehabilitation Group
Other: Daily medication — Patients will be treated with daily medication prescribed by the physician and will continue to receive the standard care from the primary care centre team.
  Arms: Standard Care Group

SUMMARY:
3R aims to increase the access of patients with chronic respiratory diseases (CRD) to pulmonary rehabilitation (PR) in Portugal. The main goals of 3R are: i) design and implement an innovative community-based PR programme; ii) assess the cost-benefit of the community-based PR programme; iii) disseminate and perform knowledge transfer about PR across the country.

PR is an evidence-based intervention for the management of CRD and offering PR has been defined as a priority by national/international organizations. However, in Portugal PR is practically inexistent (<1% of "candidate" patients have access). Currently, PR programmes are hospital-based and directed to patients with advanced disease. One of the recommendations to enhance the implementation of PR is the development on novel models of programme delivery. It is hypothesised that community-based programs, direct to patients at all grades of the disease, and involving all stakeholders (health professionals, patients, society, policy makers) may turn PR more accessible.

The plan is to implement community-based PR programs in 4 primary care centres of 2 ACES of the centre region of Portugal and assess the impact of such intervention in several domains using surrogate and patient-/family-centered outcomes. A cost-benefit analysis will be performed on acute exacerbations and healthcare utilization. Dissemination will include one conference, activities with the community, courses and an online PR toolkit. Four schools of 2 polytechnics, 2 city councils, the Health Regional Administration-Centre (ARS-Centro) and all respiratory professional and civic national associations are partners.

DETAILED DESCRIPTION:
More than 1 billion people suffer from chronic respiratory diseases worldwide and, in Europe, the total annual cost of respiratory diseases amounts to more than €380 billion. In Portugal, respiratory diseases are the 3rd leading cause of death and direct costs related to hospitalizations (in 2013 - €213 millions). Management of chronic respiratory diseases are high priorities for the National Health Service, and particularly, for the Center Health Regional Administration.

Pulmonary rehabilitation (PR) is an evidence-based intervention for the management of patients with chronic respiratory diseases (grade A). Offering PR has long been defined as a priority by several national and international organizations. Despite this firm recommendation and the knowhow on the provision of PR, in Portugal, PR is practically inexistent, with <1% of "candidate" patients having access to this standard care. Therefore, the need for a National Network on PR has been acknowledged as a priority.

It is hypothesised that community-based programmes, direct to patients at all grades of the disease, and involving all stakeholders (health professionals, patients/family, society, policy makers) may turn PR more accessible. Thus, the main goal of this project is to increase the access of patients with chronic respiratory diseases, namely COPD, to PR in the center region of Portugal and disseminate this intervention nationally.

3R aims to implement and disseminate community-based PR programs in Portugal. Specifically, it will:

1. Implement 4 community-based PR programmes (Task 1);
2. Create an online platform for clinical storage and analysis of the data collected (Task 2);
3. Perform a cost-benefit analysis of the implemented PR programmes (Task 3);
4. Create a Portuguese online PR toolkit (Task 4);
5. Promote knowledge transfer about PR (Task 5). The plan is to implement community-based PR programmes in 4 primary care centres of 2 ACES (Baixo Vouga - BV, and Baixo-Mondego - BM) of the centre region and assess the impact of such intervention in several domains. Surrogate and patient/family centered outcome measures will be used. A cost-benefit analysis will be performed on acute exacerbations and healthcare utilization and costs. Finally, dissemination and knowledge transfer of the project will be conducted through: an international conference, activities with the community, three PR courses; the development of the Portuguese online PR toolkit to support the widespread implementation of PR in Portugal and via publications.

To bring PR from bench to Portuguese common practice, 3R brings together a strong consortium composed of 4 schools of 2 Polytechnic Institutions, 2 City Councils, Health Regional Administration - Centre and all respiratory national associations (Sociedade, Portuguesa do Pulmão - SPP, RESPIRA and Fundação Portuguesa do Pulmão - FPP). This consortium involves an experienced team with complementary backgrounds and integrates students from the several institutions during all activities. It is strongly believed that jointly this multidisciplinary team has the experience and complementary skills, as well as the means, to guarantee the success and outreach of the project.

It is estimated that 73 patients will be required to detect significant differences in patients' health-related quality of life (HRQOL), based on a previous study. Stable patients with CRD and their family members will be recruited from Primary Care Centres (PCCs) of the ACES of Baixo Vouga and Baixo Mondego (ACES-BV & BM). Family doctors from PCCs will provide a list of eligible individuals. Individuals/families will be contacted and those interested will meet with researchers to receive further information about the study and sign the informed consents. Participants will be divided in two groups: experimental (EG) and control (CG). The EG will include participants/families wanting to participate in a 12-week community-based PR programme and the CG will include those willing to collaborate in data collection but not in the PR programmes (Task 1). The PR programme will include exercise training (endurance, strength and balance training) twice a week and psychoeducational sessions every two weeks performed by a multidisciplinary team.

Data will be collected at baseline, at 12 weeks (i.e., immediately post-PR), 3 and 6 months post-PR.

Data analysis will be undertaken using Statistical Package for the Social Sciences (SPSS) software and will include descriptive and inferential statistics. To analyse changes in outcome measures, data from baseline and after treatment assessments will be compared. Moreover, between groups comparisons will also be performed for baseline, after intervention and follow-ups assessments. Effect sizes for the interventions will also be calculated.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of a chronic respiratory disease
* clinically stable in the previous month
* ≥ 18 years old
* able to provide their own informed consent

Exclusion Criteria:

* cognitive impairments
* inability to understand and co-operate
* history of neoplasic /immunologic disease or acute cardiac condition or a significant cardiac, musculoskeletal, neuromuscular or psychiatric condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Health Related quality-of-life: St. George Respiratory Questionnaire | Up to 9 months
  St. George Respiratory Questionnaire (SGRQ) will be used to assess Health Related quality-of-life. The SGRQ is a comprehensive well-established 50-item questionnaire to measure health status in patients with chronic respiratory diseases. Scores can be provided for each domain and as a total score, ranging from 0 (no impairment) to 100 (worst possible health status).

SECONDARY OUTCOMES:
Change in airflow obstruction | Up to 9 months
  Forced expiratory volume in one second and forced vital capacity will be measured with a portable spirometer to assess the degree of airflow obstruction. Results will be expressed in liters and percentage of predicted. We will calculate the ratio between the forced expiratory volume in one second and the forced vital capacity.
Change in exercise capacity | Up to 9 months
  Exercise capacity will be tested in a 6-minute walk test, since it allows exercise prescription. The test results will be presented as the walked distance (meters).
Change in functionality | Up to 9 months
  Functionality will be tested with the 1-minute sit-to-stand, with the results presented as number of sit-to-stand repetitions.
Change in quadriceps muscle strength | Up to 9 months
  Quadriceps muscle strength will be measured using a handheld dynamometer (kilogram/force).
Change in biceps muscle strength | Up to 3 months
  Biceps muscle strength will be measured using a handheld dynamometer (kilogram/force).
Change in muscle cross sectional area | Up to 3 months
  Cross-sectional will be measured with ultrasound of the lower (quadriceps) and upper (biceps) limb muscles.
Change in upper limb muscle strength | Up to 9 months
  Upper limb strength will be measured with Handgrip (kg)
Change in respiratory muscle strength | Up to 3 months
  Respiratory muscle strength will be measured through a respiratory pressure meter to assess inspiratory and expiratory muscle strength (cm/H20)
Change in frequency of exacerbations | Up to 9 months
  Number of exacerbations in the previous year, healthcare utilization, such as emergency department visits or hospital admissions, in the previous year, which are related to COPD decline
Change in Healthcare utilization | Up to 9 months
  Healthcare utilization will be assessed through the number of participants that visit emergency department and the number of visits of each participant in the previous year. The number and duration of hospital admissions in the previous year will also be assessed.
Change in family adaptability/cohesion | Up to 3 months
  Family function was assessed with the family adaptability and cohesion evaluation scale (FACES-IV). The FACES-IV is a 62 items subdivided in: cohesion and flexibility dimensions, and family communication and family satisfaction scales. The cohesion and flexibility dimensions provide six family scales, two balanced scales (Balanced cohesion and balanced flexibility, with percentile scores ranging from 16 to 85) and four unbalanced scales (Disengaged, Enmeshed, Rigid and Chaotic, with percentile scores ranging from 10 to 99). The six family types (Balanced, Rigidly Cohesive, Midrange, Flexibly unbalanced, chaotically unbalanced and unbalanced) can be plotted onto the Circumplex Model. The family communications and Satisfaction scales are composed of 10 items each, with percentile scores ranging from 10 to 99. In all FACES-IV subscales higher scores indicate better family cohesion, flexibility, communication or satisfaction.
Change in balance | Up to 3 months
  Balance will be assessed with the Brief-Best tests.
Change in Physical activity | Up to 3 months
  Accelerometry will be used to assess physical activity.
Change in Physical activity | Up to 9 months
  The Brief Physical Activity questionnaire will be used to assess physical activity. It a 2 items questionnaire, with scores ranging from 0 to 8. If the sum of the two items score is above or equal 4 the subject will be considered physically active.
Change in Diaphragm excursion | Up to 3 months
  Ultrasound will be used to assess the diaphragm excursion, only volunteer from patients who agree to come to ESSUA and will be seen previously by a physician
Change in Dyspnoea | Up to 9 months
  Medical Research Council scale will be used to assess functional dyspnoea related to respiratory impairment. It is a 5-point scale, rated from 0 to 4, with higher scores denoting greater breathlessness severity.
Change in symptom's impact in patients life | Up to 9 months
  COPD Assessment Test (CAT) will be used to assess burdensome symptoms in patients' life with 8 items (cough, sputum, dyspnoea, chest tightness, capacity of exercise and home daily activities, confidence leaving home, sleep and energy levels).he scores range from 0-40, organised in 4 categories, namely <10 low impact, 10-20 medium, 21-30 high and >30 very high impact, with 5 representing the upper limit of normal in healthy non-smokers
Change in Emotional state | Up to 9 months
  Hospital Anxiety and Depression Scale will be used to assess symptoms of anxiety and depression. It is a 14 item questionnaire that can be subdivided in two subscales: anxiety and depression. Scores are provided for each subscale and range from 0 to 21, with higher scores meaning more symptoms of anxiety and depression.
Change in Fatigue symptoms | Up to 3 months
  The fatigue subscale of the Checklist of Individual Strength (CIS-20) will be used to assess fatigue.The subscale of subjective fatigue is a 8-item questionnaire, with higher scores indicating higher levels of fatigue. The total scores range from 8 to 56.
Change in Fatigue | Up to 3 months
  The Functional Assessment of Cancer Therapy - Fatigue subscale (FACIT-F) will be used to assess fatigue levels. It is multi-dimensional 13-item questionnaire assessing tiredness, weakness and difficulty in handling daily activities due to fatigue. Scores range from 0 to 52, with higher scores indicating less fatigue.
Change in cough-related quality of life: Leicester Cough Questionnaire | Up to 3 months
  Cough-related quality of life will be assessed with the Leicester Cough Questionnaire, which is a 19 items scale organised in 3 domains (physical, psychological and social). Each domain has a score ranging from 1 to 7 and the LCQ total score varies from 3 to 21. Higher scores express a better quality of life and less impact of cough.
Change in cough and sputum symptoms | Up to 3 months
  The Cough and Sputum Assessment Questionnaire (CASA-Q) will be used to assess cough and sputum symptoms, based on their reported frequency and severity, and their impact on daily activities. t is a 20-item questionnaire containing 4 domains: cough symptoms, cough impact, sputum symptoms and sputum impact. All items are rescored and summed, achieving a score ranging from 0 to 100 for each domain, with higher scores indicating fewer symptoms or less cough and sputum impact.
Digital Technology access | At baseline
  A survey asking about the use of internet and access to computers, smartphones (combination of mobile phone, web browser and computer capabilities)/tablets and cell phones (simple devices mainly for voice calls and text messages) will be used to assess digital technology access. Confidence in using these technologies will be assessed using a numerical scale from 0 (not at all confident) to 10 (completely confident).

OTHER OUTCOMES:
Change in Body Mass Index | Up to 9 months
  Patients' body mass index will be assessed in kg/m^2 based on patients' height and weight.

CONTACTS AND LOCATIONS:
Overall Officials: Alda S. Marques, PhD, Principal Investigator — School of Health Sciences of the University of Aveiro (ESSUA)
Locations (1):
- University of Aveiro, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paixao C, Rebelo P, Oliveira A, Jacome C, Cruz J, Martins V, Simao P, Marques A. Responsiveness and Minimal Clinically Important Difference of the Brief-BESTest in People With COPD After Pulmonary Rehabilitation. Phys Ther. 2021 Nov 1;101(11):pzab209. doi: 10.1093/ptj/pzab209. PMID 34499161
- [Derived] Rebelo P, Oliveira A, Andrade L, Valente C, Marques A. Minimal Clinically Important Differences for Patient-Reported Outcome Measures of Fatigue in Patients With COPD Following Pulmonary Rehabilitation. Chest. 2020 Aug;158(2):550-561. doi: 10.1016/j.chest.2020.02.045. Epub 2020 Mar 14. PMID 32184112
- [Derived] Marques A, Jacome C, Rebelo P, Paixao C, Oliveira A, Cruz J, Freitas C, Rua M, Loureiro H, Peguinho C, Marques F, Simoes A, Santos M, Martins P, Andre A, De Francesco S, Martins V, Brooks D, Simao P. Improving access to community-based pulmonary rehabilitation: 3R protocol for real-world settings with cost-benefit analysis. BMC Public Health. 2019 May 31;19(1):676. doi: 10.1186/s12889-019-7045-1. PMID 31151409